CLINICAL TRIAL: NCT02080234
Title: Combination of Gemcitabine, Oxaliplatin, and Asparaginase (GELOX) With Concurrent Involved-Field Radiation Therapy for Patients With Stage IE/IIE Extranodal Natural Killer/T-Cell Lymphoma:a Phase II Study
Brief Title: Combine GELOX With Concurrent Radiation Therapy for Patients With Stage IE/IIE ENKTL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xia Zhongjun, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GELOX1
Record Dates: First submitted 2014-03-02; First posted 2014-03-06 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Lymphoma, Extranodal NK-T-Cell
Keywords: Lymphoma, Extranodal NK-T-Cell; asparaginase; GELOX; concurrent chemoradiotherapy; sIL-2R
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — Gelox; Gemcitabine; Oxaliplatin; Asparaginase; pegaspargase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- concurrent chemoradiotherapy with GELOX (Experimental): GELOX:
  gemcitabine ：1250mg/m2 (ivdrip) on days 1, oxaliplatin :85 mg/m2 (ivdrip) on day 1, and pegaspargase : 2500 IU/m2 (intramuscular injection) on day 1.Cycle is repeated every 14 days
  IFRT
  IFRT is delivered using 6-MeV linear accelerator using 3-dimensional conformable treatment planning. The IFRT dose was 56 grays (Gy) in 28 fractions.
  the first cycle of chemotherapy was initiated on the same day of radiotherapy.
  Interventions: Drug: GELOX; Radiation: IFRT

INTERVENTIONS:
Drug: GELOX — gemcitabine ：1250mg/m2 (ivdrip) on days 1, oxaliplatin :85 mg/m2 (ivdrip) on day 1, and pegaspargase : 2500 IU/m2 (intramuscular injection) on day 1.Cycle is repeated every 14 days
  Other Names: gemcitabine; oxaliplatin; asparaginase; pegaspargase
Radiation: IFRT — IFRT is delivered using 6-MeV linear accelerator using 3-dimensional conformable treatment planning. The IFRT dose was 56 grays (Gy) in 28 fractions

SUMMARY:
To evaluate the efficacy and safety of first-line gemcitabine, oxaliplatin, and asparaginase (GELOX) with concurrent involved-field radiation therapy for patients in newly diagnosed stage IE/IIE ENKTL.

DETAILED DESCRIPTION:
1. Patients

   * All patients should sign a written informed consent form before enrollment, and the study should be approved by the Sun Yat-sen University Cancer Center Ethics Board.
   * Baseline of patients: Computed tomography (CT) scans of the chest, abdomen, and pelvis, magnetic resonance imaging studies of the head and neck, and bilateral bone marrow aspiration or biopsy. Positron emission tomography-CT scans (optional). Epstein-Barr virus (E B V) DNA blood levels, titer of EBV antibody (EA-IgA, VCA-IgA), β2-micro globulin (β2-MG) and soluble CD 25 (sCD 25) in the serum.
   * Recheck before and after every course: Epstein-Barr virus (EBV) DNA blood levels, titer of EBV antibody (EA-IgA, VCA-IgA), β2-micro globulin (β2-MG) and soluble CD 25 (sCD25) in the serum.
   * Recheck every two course: Computed tomography (CT) scans of the chest, abdomen, and pelvis, magnetic resonance imaging studies of the head and neck, and bilateral bone marrow aspiration or biopsy. Positron emission tomography-CT scans (optional)
2. Treatment Protocol - The GELOX regimen consist of the following drugs: gemcitabine ：1250 mg/ m2 on days 1,ivdrip oxaliplatin ：85 mg/m2 on day 1, ivdrip pegaspargase : 2500 IU/m 2 daily on day 1,intramuscular The treatment cycle was repeated every 14 days.

   * IFRT was delivered using 6-MeV linear accelerator using 3-dimensional conformable treatment planning. The IFRT dose was 56 grays (Gy) in 28 fractions, we define the clinical target volume of limited stage IE disease as the bilateral nasal cavity, bilateral ethmoid sinuses, and ipsilateral maxillary sinus; and the clinical target volume would extend to involved tissues for patients who had extensive stage IE disease. For patients who had stage IIE disease, the clinical target volume also, included the bilateral cervical lymph node area.

     * Disease Progression during the treatment should be treated with second-line therapy.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed ENKTL
* age:18-69years
* Ann Arbor stage IE,or stage IIE with cervical lymph node involvement
* at lease one measurable lesion
* receive no chemotherapy or radiotherapy before
* Eastern CooperativeOncology Group performance status of 0 to 2.
* Adequate hematologic function (eg, white blood cell ≥ 3×10e9/l,neutrophils count ≥1.5×10e9/L, and platelet count≥ 100×10e9/L),renal function (eg, serum creatinine≤1.5 mg/dL and creatinine clearance ≥50 mL minute), and hepatic function (e.g, total bilirubin≤ 2 times the upper limit of normal and aspartate and alanine transaminase levels ≤ 3 times the upper limit of normal)

Exclusion Criteria:

* mismatch the inclusion criteria
* systematic central nervous system involvement, previous or concomitant malignancies and any coexisting medical problems that could cause poor compliance with the study protocol.
* primary lesion not from the upper respiratory

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
complete remission rate | every 4 weeks,up to completion of treatment(approximately 6 months)
  1.The criteria for the efficacy evaluation (overall response rate and complete remission) of the regimen is according to the following article.
  Cheson BD, Horning SJ, Coiffier B, et al. Report of an international workshop to standardize response criteria for non-Hodgkin's lymphomas. NCI Sponsored International Working Group. J Clin Oncol. 1999;17:1244.

SECONDARY OUTCOMES:
progression free survival | up to end of follow-up-phase (approximately 3 years)
  progression free survival(PFS): time from the date of enrollment to date of disease progression, or death of any cause, or date of lost follow-up, whichever comes first
overall survival | up to end of follow-up-phase (approximately 3 years)
  overall survival (OS): time from the date of enrollment to date of death from any cause, or date of lost follow-up, whichever comes first.
safety | up to end of follow-up-phase (approximately 3 years)
  including hematological safety and non-hematological safety.All the adverse events will be classified according to Common Terminology Criteria for Adverse Events v3.0 (CTCAE)

OTHER OUTCOMES:
Epstein-Barr virus(EBV) DNA copies | Time Frame: every 3 weeks,up to completion of treatment(approximately 6 months)
Plasma β2-microglobulin | every 3 weeks,up to completion of treatment(approximately 6 months)
serum sIL-2R level | every 3 weeks,up to completion of treatment(approximately 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: ZhongJun Xia, MD/PHD, Principal Investigator — Department of Hematological Oncology, Sun Yat-sen University Cancer Center; State Key Laboratory of Oncology in South China,
Locations (1):
- Sun Yat-sen University Cancer Center; State Key Laboratory of Oncology in South China,, Guangzhou, Guangdong, China